CLINICAL TRIAL: NCT04765020
Title: Effects of a Physical Activity Program on Cardiorespiratory Fitness in Children and Adolescents FolloWing Acute CancER Treatment: a Randomized Controlled Trial
Brief Title: Cardiorespiratory Fitness in Children and Adolescents After Cancer Treatment.
Acronym: POWER
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Helios Hospital Krefeld (Unknown); Oslo Centre for Biostatistics and Epidemiology (Unknown); University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Miriam Götte, Dr. rer. medic. Miriam Götte, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HCRI ID 2020-0250
Record Dates: First submitted 2021-01-26; First posted 2021-02-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: All Types of Pediatric Cancer
Keywords: exercise; cardiorespiratory fitness; pediatric oncology; child health; physical activity; immune function
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): 12 weeks moderate to high-intensity exercise program
  Interventions: Behavioral: Experimental: moderate to high-intensity exercise
- Control group (No Intervention): exercise recommendations

INTERVENTIONS:
Behavioral: Experimental: moderate to high-intensity exercise — Four parts:
  1. Initial consultation with recommendations for general physical activity, brochure with exercise recommendations
  2. Once per week multi-modal group-based exercise (endurance, strength, mobility, coordination)
  3. Once per week supervised multi-modal individual training session (endurance, strength, mobility, coordination). Intensity: 60-80% of max. HR
  4. Activity trackers with individual movement goals that will be adjusted every two weeks
  Other Names: 12-week, partially supervised exercise program; general exericse recommendationy
  Arms: Intervention group

SUMMARY:
The POWER-study is a two-arm exercise intervention study for pediatric patients following acute cancer treatment. This clinical trial will investigate the effects of a 12-week moderate to high-intensity exercise program on cardiorespiratory fitness in children and adolescents beginning 6 weeks after completion of acute cancer treatment.

DETAILED DESCRIPTION:
The main objective of the POWER study is to investigate the effects of a 12-week moderate to high-intensity, partially supervised exercise program on cardiorespiratory fitness (VO2peak) in children and adolescents who have completed acute cancer treatment. This randomized controlled trial will include n=56 patients. Patients will be randomly assigned to the intervention or the control group. Patients in the intervention group will perform two supervised exercise sessions per week, one personal training session and one group-based training session. During an initial consultation, both groups receive recommendations for individual physical activity goals and a brochure with exercise recommendations as well as a fitness tracker to monitor their daily physical activity. Only the intervention group will receive daily activity targets, which will be adjusted on a regular basis. The study starts 6 weeks after completion of the patient's acute cancer treatment.

Secondary aims of this interventional study are to evaluate additional performance markers, including muscle strength, functional mobility, balance, body composition and patient-reported outcomes including QoL, fatigue, and cognitive function as well as blood markers to evaluate changes in metabolic, immune, and heart health.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 7 and 23 years of age
* Completion of acute cancer treatment and receiving follow-up care in Krefeld (Helios Hospital Krefeld)
* 6 weeks post cancer-treatment
* Signed informed consent (Parents and Patient)

Exclusion Criteria:

* <7 years of age, >23 years of age
* Medical condition that limits participation in one of the study arms
* Inability to follow the training-protocol
* Inability to carry out the spiroergometry on a cycle ergometer

Ages: 7 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in maximal oxygen uptake (VO2peak, ml/kg/min) from Baseline to T1 (end of intervention/12-weeks post randomization) between the two study groups, assessed in a maximal incremental exercise test (CPET) on a bicycle ergometer. | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  CPET is performed on an electronically braked cycle ergometer (Ergoline ergoselect 150 P) following the GDPK-Ergometry-Protocol). Ventilation and gas exchange data are determined breath-by-breath (Geratherm Respiratory Ergostik). VO2 peak is defined as the highest mean over 60 s and expressed on milliliters/kilogram/minute (ml/kg/min).

SECONDARY OUTCOMES:
Adverse events | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
Muscle strength | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  Change in maximal muscle strength (CITEC handheld dynamometer; expressed in Newton), balance (single leg stance; expressed in seconds), functional mobility (TUG 3m; expressed in seconds), and body composition (Data Input Nutribox) between both study arms from T0 to T1, T0 to T2 and T1 to T2
Functional mobility | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  Time (in sec) to complete the Timed Up and Go Test (TUG). The participants perform one test trial. The time of standing up, walking at a safe and comfortable pace to a mark 3 meters away from them, returning to the chair and sitting back down is recorded.
Static Balance | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  Single leg stance on a wooden bar, adapted by the MOON test, number of times the ground is touched during a one-minute test procedure
Body Composition | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  Body composition is assessed by bioimpedance analysis. Whole body resistance and reactance are measured using the BIA device Data Input Nutribox.
Change in level of physical activity | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  3. Change in level of physical activity (questionnaire and activity monitor) between both study arms at T1 and T2 and intra-individually
Change in Quality of Life | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  (PedsQL - Pediatric Quality of Life Inventory), change in Fatigue (Multidimensional Fatigue Inventory) and cognitive function (Ravens Progressive; WISC V - subtest memory; TAP ) between both study arms at T1 and T2 and intra-individually
Changes in serum markers | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  CRP, BDNF, Insulin, Glukose, Adiponectin, Leptin, IL-1 beta, IL-2, IL-4, IL-6, IL-7, IL-8, IL-10, IL-15, IL 17a, TNF alpha, CRP, BDNF, IGF 1, MIF (macrophage migration inhibiting factor), IFN gamma, Troponin, NT-pro-BNP, between both study arms at T1 and T2 and intra-individually
Changes in Echocardiography markers | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  M-Mode-Parameter
Changes in Echocardiography markers | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  Left ventricle end diastolic volume (LVEDV) in ml/m²
Changes in Echocardiography markers | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  Ejection Fraction (EF) in %
Changes in Echocardiography markers | At Baseline T0: 6 weeks following acute cancer treatment, T1: after 12 weeks of intervention, T2 (Follow up): after 12 weeks after end of intervention = 24 weeks after study inclusion
  Tricuspid Annular Plane Systolic Excursion (TAPSE) in Millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Götte, Phd, Principal Investigator — University Hospital, Essen
Locations (1):
- Helios Klinik Krefeld, Krefeld, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol